CLINICAL TRIAL: NCT02539316
Title: Pilot Study: Hepatoprotective Role of SMOFlipid® Used in Short-term Parenteral Nutrition in an Onco-Hematology Pediatric Population
Acronym: SMOFPILOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-PP-03
Record Dates: First submitted 2015-08-11; First posted 2015-09-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Dietary and Nutritional Therapies
Keywords: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia | interventions — SMOFlipid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Médialipides (Active Comparator): parenteral nutrition by Médialipides (dosage form depending child's weight as recommended by the SPC)
  Interventions: Drug: Médialipides
- SmofLIPID (Experimental): parenteral nutrition by Smoflipid (dosage form depending child's weight as recommended by the SPC)
  Interventions: Drug: Smoflipid

INTERVENTIONS:
Drug: Smoflipid
  Arms: SmofLIPID
Drug: Médialipides
  Arms: Médialipides

SUMMARY:
Parenteral nutrition (PN) is part of supportive care in oncology Pediatric when the patient's nutritional status justifies it and enteral is impossible. In the literature, hepatotoxicity, cholestasis type, standard emulsions of soy oil-based (type Médialipide®) is described in the context of a long-term PN especially in premature infants. It results in an increase in gammaGT. The most recent use of lipid emulsions containing Omega 3 (Smoflipid), was studied in the adult population and in the preterm in the PN on short and long, with the finding of a hepatoprotection. Investigators do not find a single retrospective study about it in Pediatric Onco-Hematology. No prospective studies have been performed in the population of Onco-Hematology. The objective of this study is to evaluate the impact of the use of SMOFlipid® in parenteral nutrition on early occurrence of cholestasis compared with Médialipides in a short-term use of parenteral nutrition in an Onco-Hematology pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years
* Solid Tumors
* hematological malignancies
* Requiring parenteral nutrition during at least 5 days
* With a central catheter
* With a normal hepatic function test

Exclusion Criteria:

* Liver function tests disrupted
* Patient with a tumor or liver metastases
* Patient with against-indication to the use of lipid

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
dosage of γGT in UI/l | Baseline
  to evaluate the impact of the use of SMOFlipid® in parenteral nutrition on early occurrence of cholestasis compared with Médialipides in a short-term use of parenteral nutrition in an Onco-Hematology pediatric population.
dosage of γGT in UI/l | at day 5
dosage of γGT in UI/l | 7 days after the end of parenteral nutrition

SECONDARY OUTCOMES:
asat, alat, PAL, LDH, total bilirubin CRP | Baseline
asat, alat, PAL, LDH, total bilirubin CRP | at day 5
asat, alat, PAL, LDH, total bilirubin CRP | 7 days after the end of parenteral nutrition
Triglycerids Digestive tolerance (vomiting) | Baseline
Triglycerids Digestive tolerance (vomiting) | at day 5
Triglycerids Digestive tolerance (vomiting) | 7 days after the end of parenteral nutrition
Infectious episodes (numbers, duration) | Baseline
Infectious episodes (numbers, duration) | at day 5
Infectious episodes (numbers, duration) | 7 days after the end of parenteral nutrition
Nutritionnal status | Baseline
  (Albumin, weight, BMI)
Nutritionnal status | at day 5
  (Albumin, weight, BMI)
Nutritionnal status | 7 days after the end of parenteral nutrition
  (Albumin, weight, BMI)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de l'Archet - CHU de Nice, Nice, France